CLINICAL TRIAL: NCT00000124
Title: Collaborative Ocular Melanoma Study (COMS)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Eye Institute (NEI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NEI-23
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2006-06-02 (Estimated); Status verified 2002-06

CONDITIONS: Choroid Neoplasms; Uveitis
Keywords: Choroidal Melanoma; Ocular Melanoma
MeSH Terms: conditions — Choroid Neoplasms; Uveitis; Uveal Melanoma | interventions — Brachytherapy; Eye Enucleation

INTERVENTIONS:
Procedure: Brachytherapy
Procedure: Eye Removal

SUMMARY:
To evaluate therapeutic interventions for patients who have choroidal melanoma, the most common primary eye cancer affecting adults, and to assess the potential life-preserving as well as sight-preserving role of radiation therapy.

To determine which of two standard treatments, removal of the eye or brachytherapy, is more likely to prolong survival of eligible patients with medium-sized choroidal melanoma.

To determine whether preoperative radiation prolongs life for patients whose eyes with large choroidal melanoma are enucleated.

DETAILED DESCRIPTION:
For more than 100 years, removal of the eye (enucleation) has been the standard treatment for choroidal melanoma. Before the COMS was initiated in 1986, interest in radiation therapy had increased because of the potential for saving the eye and perhaps some vision. However, the merits of radiation with respect to prolonging patient survival were unknown. The best data from nonrandomized studies suggested that there was no difference in length of remaining life between patients treated with radiation and those whose eyes were enucleated. Thus, it was appropriate and necessary to conduct a randomized, controlled clinical trial in which a large number of patients would be followed for many years in order to compare enucleation and radiation with respect to relative success in prolonging survival of choroidal melanoma patients.

The Collaborative Ocular Melanoma Study (COMS) is a set of long-term, multicenter, randomized controlled trials. In the trial for patients with tumors of medium size, enucleation and irradiation with an iodine-125 episcleral plaque are compared on the basis of length of remaining life. All randomized patients will be followed for 5 to 15 years or until death. For patients randomly assigned to enucleation, the eye was removed following a standard procedure. For patients assigned to plaque irradiation, the margins of the tumor were located and the dimensions of the tumor were measured by the ophthalmic surgeon. A gold plaque with a plastic seed carrier that contained the proper dosage and configuration of radioactive iodine seeds was sutured to the outside (sclera) of the eye over the base of the tumor. This procedure made possible the delivery of a high dose of radiation to a very localized area (85 Gy [TG-43] to the tumor apex). The plaque typically was removed from the eye after three to seven days. Enrollment was completed in this trial in July 1998 with 1,317 patients enrolled. Clinical follow-up of patients will end in July 2003.

In the COMS trial of preoperative radiation, patients with large tumors were randomized to enucleation alone or to enucleation preceded by 20 Gy of external beam radiation. The two randomly assigned groups of patients were followed for at least five years or until death and have been compared on the basis of length of remaining life and other outcomes. Enrollment in this trial was completed in December 1994, with 1,003 patients enrolled. Clinical follow-up of all patients in this trial ended in July 2000.

Accrual to a nonrandomized pilot study to assess the feasibility of a randomized trial for small tumors was halted in 1989. Additional followup of those 204 patients was carried out from 1994 to 1996.

The COMS is conducted in 43 clinical centers located in major population areas of the United States and Canada. Six resource centers participate and have major roles in quality assurance for the study. Information gathered and analyzed includes time to death from all causes, time to death from cancer (whether metastatic choroidal melanoma or not), diagnosis of other tumors, complications of radiation, and changes in visual acuity. A parallel study of quality of life for patients enrolled in the trial of radioactive plaque was initiated in January 1995. From November 1986 through July 1998, 8,712 patients with choroidal melanoma of all sizes were screened for eligibility for a COMS clinical trial.

ELIGIBILITY:
Men and women eligible for the study must be age 21 or older, have primary choroidal melanoma in only one eye, and have no evidence of metastatic disease. Accurate estimation of tumor thickness by echography must also be possible.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1986-11

REFERENCES:
- [Background] Byrne SF, Marsh MJ, Boldt HC, Green RL, Johnson RN, Wilson DJ. Consistency of observations from echograms made centrally in the Collaborative Ocular Melanoma Study COMS Report No. 13. Ophthalmic Epidemiol. 2002 Feb;9(1):11-27. doi: 10.1076/opep.9.1.11.1719. PMID 11815892
- [Background] Collaborative Ocular Melanoma Study Group. Sociodemographic and clinical predictors of participation in two randomized trials: findings from the Collaborative Ocular Melanoma Study COMS report no. 7. Control Clin Trials. 2001 Oct;22(5):526-37. doi: 10.1016/s0197-2456(01)00157-x. PMID 11578786
- [Background] Moy CS, Albert DM, Diener-West M, McCaffrey LD, Scully RE, Willson JK; Collaborative Ocular Melanoma Study Group, prepared by COMS Mortality Coding Committee. Cause-specific mortality coding. methods in the collaborative ocular melanoma study coms report no. 14. Control Clin Trials. 2001 Jun;22(3):248-62. doi: 10.1016/s0197-2456(01)00113-1. PMID 11384789
- [Background] Collaborative Ocular Melanoma Study Group.. Assessment of metastatic disease status at death in 435 patients with large choroidal melanoma in the Collaborative Ocular Melanoma Study (COMS): COMS report no. 15. Arch Ophthalmol. 2001 May;119(5):670-6. doi: 10.1001/archopht.119.5.670. PMID 11346394
- [Background] Melia BM, Abramson DH, Albert DM, Boldt HC, Earle JD, Hanson WF, Montague P, Moy CS, Schachat AP, Simpson ER, Straatsma BR, Vine AK, Weingeist TA; Collaborative Ocular Melanoma Study Group. Collaborative ocular melanoma study (COMS) randomized trial of I-125 brachytherapy for medium choroidal melanoma. I. Visual acuity after 3 years COMS report no. 16. Ophthalmology. 2001 Feb;108(2):348-66. doi: 10.1016/s0161-6420(00)00526-1. PMID 11158813
- [Background] Echography (Ultrasound) Procedures for the Collaborative Ocular Melanoma Study (COMS), Report no. 12, Part II. J Ophthalmic Nurs Technol. 1999 Sep-Oct;18(5):219-32. No abstract available. PMID 10847049
- [Background] Echography (ultrasound) procedures for the Collaborative Ocular Melanoma Study (COMS), Report no. 12, Part I. J Ophthalmic Nurs Technol. 1999 Jul-Aug;18(4):143-9. No abstract available. PMID 10847038
- [Background] Quality of life assessment in the collaborative ocular melanoma study: design and methods. COMS-QOLS Report No. 1. COMS Quality of Life Study Group. Ophthalmic Epidemiol. 1999 Mar;6(1):5-17. doi: 10.1076/opep.6.1.5.1565. PMID 10384680
- [Background] The Collaborative Ocular Melanoma Study (COMS) randomized trial of pre-enucleation radiation of large choroidal melanoma III: local complications and observations following enucleation COMS report no. 11. Am J Ophthalmol. 1998 Sep;126(3):362-72. doi: 10.1016/s0002-9394(98)00091-9. PMID 9744369
- [Background] The Collaborative Ocular Melanoma Study (COMS) randomized trial of pre-enucleation radiation of large choroidal melanoma II: initial mortality findings. COMS report no. 10. Am J Ophthalmol. 1998 Jun;125(6):779-96. doi: 10.1016/s0002-9394(98)00039-7. PMID 9645716
- [Background] The Collaborative Ocular Melanoma Study (COMS) randomized trial of pre-enucleation radiation of large choroidal melanoma I: characteristics of patients enrolled and not enrolled. COMS report no. 9. Am J Ophthalmol. 1998 Jun;125(6):767-78. doi: 10.1016/s0002-9394(98)00038-5. PMID 9645715
- [Background] Histopathologic characteristics of uveal melanomas in eyes enucleated from the Collaborative Ocular Melanoma Study. COMS report no. 6. Am J Ophthalmol. 1998 Jun;125(6):745-66. doi: 10.1016/s0002-9394(98)00040-3. PMID 9645714
- [Background] Factors predictive of growth and treatment of small choroidal melanoma: COMS Report No. 5. The Collaborative Ocular Melanoma Study Group. Arch Ophthalmol. 1997 Dec;115(12):1537-44. doi: 10.1001/archopht.1997.01100160707007. PMID 9400787
- [Background] Grossniklaus HE, Albert DM, Green WR, Conway BP, Hovland KR. Clear cell differentiation in choroidal melanoma. COMS report no. 8. Collaborative Ocular Melanoma Study Group. Arch Ophthalmol. 1997 Jul;115(7):894-8. doi: 10.1001/archopht.1997.01100160064010. PMID 9230830
- [Background] Mortality in patients with small choroidal melanoma. COMS report no. 4. The Collaborative Ocular Melanoma Study Group. Arch Ophthalmol. 1997 Jul;115(7):886-93. PMID 9230829
- [Background] Wells CG, Bradford RH, Fish GE, Straatsma BR, Hawkins BS. Choroidal melanomas in American Indians. COMS Group. Collaborative Ocular Melanoma Study. Arch Ophthalmol. 1996 Aug;114(8):1017-8. doi: 10.1001/archopht.1996.01100140225024. No abstract available. PMID 8694711
- [Background] Design and methods of a clinical trial for a rare condition: the Collaborative Ocular Melanoma Study. COMS Report No. 3. Control Clin Trials. 1993 Oct;14(5):362-91. doi: 10.1016/0197-2456(93)90052-f. PMID 8222668
- [Background] Accuracy of diagnosis of choroidal melanomas in the Collaborative Ocular Melanoma Study. COMS report no. 1. Arch Ophthalmol. 1990 Sep;108(9):1268-73. doi: 10.1001/archopht.1990.01070110084030. PMID 2205183
- [Background] Earle J, Kline RW, Robertson DM. Selection of iodine 125 for the Collaborative Ocular Melanoma Study. Arch Ophthalmol. 1987 Jun;105(6):763-4. doi: 10.1001/archopht.1987.01060060049030. No abstract available. PMID 3579705
- [Background] Diener-West M, Earle JD, Fine SL, Hawkins BS, Moy CS, Reynolds SM, Schachat AP, Straatsma BR; Collaborative Ocular Melanoma Study Group. The COMS randomized trial of iodine 125 brachytherapy for choroidal melanoma, III: initial mortality findings. COMS Report No. 18. Arch Ophthalmol. 2001 Jul;119(7):969-82. doi: 10.1001/archopht.119.7.969. PMID 11448319
- [Background] Diener-West M, Earle JD, Fine SL, Hawkins BS, Moy CS, Reynolds SM, Schachat AP, Straatsma BR; Collaborative Ocular Melanoma Study Group. The COMS randomized trial of iodine 125 brachytherapy for choroidal melanoma, II: characteristics of patients enrolled and not enrolled. COMS Report No. 17. Arch Ophthalmol. 2001 Jul;119(7):951-65. doi: 10.1001/archopht.119.7.951. PMID 11448318
- [Derived] Boldt HC, Melia BM, Liu JC, Reynolds SM; Collaborative Ocular Melanoma Study Group. I-125 brachytherapy for choroidal melanoma photographic and angiographic abnormalities: the Collaborative Ocular Melanoma Study: COMS Report No. 30. Ophthalmology. 2009 Jan;116(1):106-115.e1. doi: 10.1016/j.ophtha.2008.10.013. PMID 19118701
- [Derived] Fine SL, Hawkins BS. The investigators' perspective on the collaborative ocular melanoma study. Arch Ophthalmol. 2007 Jul;125(7):968-71. doi: 10.1001/archopht.125.7.968. No abstract available. PMID 17620582
- [Derived] Collaborative Ocular Melanoma Study Group. Incidence of cataract and outcomes after cataract surgery in the first 5 years after iodine 125 brachytherapy in the Collaborative Ocular Melanoma Study: COMS Report No. 27. Ophthalmology. 2007 Jul;114(7):1363-71. doi: 10.1016/j.ophtha.2006.10.039. Epub 2007 Mar 6. PMID 17337065
- [Derived] Collaborative Ocular Melanoma Study Group. The COMS randomized trial of iodine 125 brachytherapy for choroidal melanoma: V. Twelve-year mortality rates and prognostic factors: COMS report No. 28. Arch Ophthalmol. 2006 Dec;124(12):1684-93. doi: 10.1001/archopht.124.12.1684. PMID 17159027